CLINICAL TRIAL: NCT04245501
Title: Threat Interpretation Bias as Cognitive Marker and Treatment Target in Pediatric Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Rozenman, Assistant Professor, Department of Psychology, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R61MH121552-01 (NIH); 1R61MH121552 (NIH)
Record Dates: First submitted 2020-01-12; First posted 2020-01-29 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders
Keywords: Child; Adolescent; Pediatric; Youth; Anxiety; Separation anxiety; Social phobia; Social anxiety; Generalized anxiety; Interpretation bias; Cognitive bias; Cognitive bias modification; Interpretation bias modification; Randomized controlled trial; Threat bias; Threat interpretation; Intervention; Randomized; Cognitive training; National Institute of Mental Health; Personalized
MeSH Terms: conditions — Anxiety Disorders; Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Eligible youth will be randomly assigned to receive either 16 sessions of a personalized cognitive bias modification for interpretation bias (CBM-I) intervention or a computerized interpretation control condition (ICC). Regardless of randomization, participants will complete 16 sessions of their assigned condition within 4 weeks (1 in-lab training per week, and 3 at-home trainings per week).
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blind to condition. Unblinding occurs following all post-intervention assessment (i.e., after 16 CBM-I or ICC sessions).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification for Interpretations (CBM-I) (Experimental): Computerized 16-session intervention aimed at reducing interpretation bias. In this study, CBM-I is personalized to youth anxiety symptoms. During CBM-I sessions, youth indicate whether word-sentence pairs are related, and are provided with feedback aimed to reduce bias.
  Interventions: Other: Cognitive Bias Modification for Interpretations (CBM-I)
- Interpretation Control Condition (ICC) (Placebo Comparator): Computerized 16-session intervention that is not believed to significantly modify bias. In this study, youth see stimuli personalized to their anxiety symptoms. During ICC sessions, youth see word-sentence pairs and are required to indicate whether word and sentence are related, but are not provided with feedback that aims to "train" a reduction in interpretation bias.
  Interventions: Other: Interpretation Control Condition (ICC)

INTERVENTIONS:
Other: Cognitive Bias Modification for Interpretations (CBM-I) — Computerized intervention in which youth see word-sentence pairs personalized to their anxiety symptoms, and indicate whether these are related. Youth receive feedback aimed to reduce interpretation bias.
  Other Names: Interpretation bias modification; Interpretation training
  Arms: Cognitive Bias Modification for Interpretations (CBM-I)
Other: Interpretation Control Condition (ICC) — Computerized control condition in which youth see word-sentence pairs personalized to their anxiety symptoms. Youth indicate whether these are related, but are not provided with feedback that aims to "train" a reduction in interpretation bias.
  Arms: Interpretation Control Condition (ICC)

SUMMARY:
Anxiety is the most common mental health problem in children and adolescents. This two-phased study will test the effects of an experimental computerized intervention aimed at reducing threat-based thinking (i.e., interpretation bias) in anxious youth. Participants in both the R61 (N=46) and R33 (N=72) trials will be youth ages 10 to 17 with a primary anxiety disorder (Separation, Social, Generalized). In the R61 trial, youth will be randomly assigned to receive 16 sessions over 4 weeks of either a personalized cognitive bias modification program for interpretation bias (CBM-I) or a computerized control condition (ICC). If CBM-I reduces interpretation bias significantly more than the ICC, the R33 trial will commence. In the R33, youth will be randomly assigned to either CBM-I or an equal amount of time in a cognitive restructuring intervention, which also aims to reduce threat-based thinking in anxiety. Please note that only the R61 phase of the trial has been completed and currently this record summary only reflects the R61 phase.

DETAILED DESCRIPTION:
Anxiety is the most common mental health problem in youth, affecting one in four children and adolescents. Unfortunately, evidence-based treatments (pharmacotherapy, cognitive-behavioral therapy) are costly, not widely available, and ineffective for a substantial proportion of youth. In response, experts have called for novel treatments that directly target mechanisms underlying youth anxiety while simultaneously addressing barriers to care (i.e., cost, accessibility). One such promising mechanism is interpretation bias - the inaccurate interpretation of threat from ambiguity. The investigators have previously demonstrated that interpretation bias occurs in over 90% of anxious youth, is predictive of anxiety severity in clinical samples of youth, and differentiates between anxious and non-anxious youth. These data indicate that interpretation bias may be a ubiquitous phenomenon underlying anxiety expression in children and adolescents and therefore may be an ideal intervention target. Cognitive bias modification for interpretation bias (CBM-I) is a computerized intervention that attempts to reduce anxiety by directly modifying interpretation bias. CBM-I has demonstrated preliminary efficacy for reducing anxiety symptoms in adults. Yet extant CBM-I data in anxious youth are sparse, with little work addressing whether CBM-I significantly reduces interpretation bias, and whether this in turn reduces anxiety symptoms, as well as the dose necessary to reduce both bias and anxiety. This two-phased study tests personalized CBM-I in youth ages 10 to 17 who meet diagnostic criteria for a primary anxiety disorder (Separation, Social, Generalized). In the R61 Phase (N=46), a randomized clinical trial (RCT) examines whether CBM-I personalized to youth anxiety symptoms significantly reduces interpretation bias compared to a computerized interpretation control condition (ICC). The interpretation target will be measured at multiple time points (4, 8, 12, 16 sessions) to identify the optimal dose for reduction in interpretation bias. If the R61 trial results indicate that CBM-I outperforms ICC on interpretation bias reduction, the R33 phase will commence. In the R33 Phase, an RCT (N=72) will validate whether CBM-I significantly reduces interpretation bias, and conducts a mechanism test (i.e., does bias reduction precede and predict anxiety reduction?), by comparing CBM-I to cognitive restructuring, a clinically relevant psychosocial intervention that also targets anxious cognition. Please note that only the R61 phase of the trial has been completed and currently this record summary only reflects the R61 phase. If the R33 phase is funded, it will be registered as a separate NCT.

ELIGIBILITY:
Inclusion Criteria:

* youth aged 10 to 17
* diagnosed at study baseline with a primary "big three" anxiety disorder (Separation, Social, Generalized)
* standard score greater than or equal to 85 on the Wide Range Achievement Test - Word Reading Subtest (to ensure ability to read stimuli during interpretation bias assessment and CBM-I/ICC), and estimated IQ standard score of at least 80 on the Wechsler Abbreviated Scale of Intelligence
* youth and consenting parent/legal guardian speak sufficient English to complete consent/assent and study procedures
* no concurrent psychosocial services during study participation to reduce likelihood that other interventions are responsible for change in primary or secondary outcomes
* no psychotropic medications with no plans to start medications during study, or six weeks stable on SSRI or psychostimulant medication and dose with no plans to change medication/dose during study

Exclusion Criteria:

* severe anxiety indicting that youth requires higher level of care (e.g., intensive treatment such as psychiatric hospitalization), significant diagnostic comorbidity (e.g., presence of psychosis or significant mood disorder), or another primary diagnosis that warrants alternate intervention
* significant uncorrected vision impairment (e.g., uncorrected blindness) that precludes participation in CBM-I/ICC
* safety concerns due to recent or acute suicidality with plan, intent, and/or attempt that warrants alternate intervention

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Rozenman, Ph.D., Principal Investigator — University of Denver
Locations (1):
- BRAVE Lab, Department of Psychology, University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data resulting from this project will be de-identified and uploaded in a timely manner to the National Database for Clinical Trials Related to Mental Illness, including de-identified youth demographic and clinical characteristics, and summary scores from outcome measures, along with a data dictionary that provides variable definitions, value labels, and scoring of measures. The study protocol and dataset may be made available to other investigators based on successful completion of a data request form, following the conclusion of this study and publication of primary outcome papers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available following conclusion of the study and publication of primary outcome papers.
Access Criteria: Researchers will be required to complete a request form that includes: research identifying information and institutional affiliation, description of research objectives, and IRB approval. Completed request forms will be reviewed by the PI and Co-Is to ensure that the research request will not duplicate work being conducted by the study team. The requesting researcher must provide signed data sharing agreements from all users on their team outlining the details of how information will be kept secure, consistent with NIMH and University of Denver data sharing guidelines. Requesting researchers will also provide the University of Denver's IRB with an IRB approval from their institution. The data will only be released after the proposed study has been completed and primary outcomes have been accepted for publication.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that youth were enrolled in the study and their caregiver completed questionnaires and diagnostic interviews about the youth (not about themselves as caregivers/adults). As such, youth were the only true participants in the study (i.e., this was not dyad recruitment and caregivers did not participate as study participants but as additional reporters on the youths' symptoms as is typical in clinical anxiety trials with child and adolescent participants).
Period: Overall Study
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Started | 25 | 25
Completed | 23 (Two siblings dropped treatment after training session 2 due to one of the siblings' medical hospitalization for an unrelated, congenital medical problem.) | 24 (One youth was randomized but we learned at training session 1 that they had been receiving CBT and were therefore ineligible to continue in study.)
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — ineligible participant unknowingly enrolled | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.76 (1.64) | 12.20 (1.80) | 12.48 (1.73)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Youth self-identified gender: Female | 15 | 15 | 30
  Youth self-identified gender: Male | 9 | 8 | 17
  Youth self-identified gender: Non-binary | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 23 | 20 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 19 | 42
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Linguistic Interpretation Bias as Assessed by the Word-sentence Association Paradigm for Youth (WSAP-Y)
Description: The WSAP-Y is a computerized assessment of interpretation bias in which youth indicate whether word-sentence pairings are related. This measure provides information about the degree to which youth evidence interpretation bias, as well as a behavioral (reaction time) index for bias endorsement. For the primary outcome of percent threat interpretations endorsed, the possible range is 0 (zero) to 100%. Higher percentage indicates more threat interpretation bias (i.e., the youth endorsed a higher proportion of threat words as related to amiguous sentences); lower scores indicate lower threat interpretation bias. Greater decrease in the percent of threat interpretations endorsed and lower absolute scores indicate "better" outcome (i.e., more reduction in threat interpretation bias; less interpretation bias overall).
Time Frame: 6 weeks; post-intervention time point
Population: The WSAP-Y analysis was a between-groups analysis of interpretation bias as measured by percent threat interpretations endorsed during the task. The outcome measures data below provides the percent threat interpretations endorsed at the post-treatment (6 weeks) endpoint, and does not reflect the complex linear, quadratic, and piecewise models of change for analyses in Aims 1 and 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Number analyzed (Participants) | 25 | 25
score on a scale | 19.77 (19.48) | 47.40 (13.52)

2. Primary Outcome: Change in Visual Interpretation Bias as Assessed by the Ambiguous Faces Task
Description: Youth view faces portraying neutral expressions or subtle emotional expressions (i.e., morphed faces ranging in intensity of emotional valence). Youth categorization of faces as neutral or threatening provides their sensitivity and bias for reporting presence of threat. The criterion mean value in outcomes below reflects a score from -1 to 1, with higher negative numbers reflecting greater bias toward angry faces, and higher positive values approaching one reflecting a bias toward happy faces. Theoretically, higher positive values indicate "better" outcome such that youth have more positive bias toward facial stimuli. H
Time Frame: 6 weeks; post-intervention time point
Population: The faces analysis was a between-groups analysis of interpretation bias as measured using signal detection theory. The analysis was a between-groups analysis of interpretation bias for detecting anger versus happy faces. The outcome measures data below provides the measure endorsed at the post-treatment (6 weeks) endpoint, and does not reflect the complex linear, quadratic, and piecewise models of change for analyses in Aims 1 and 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Number analyzed (Participants) | 25 | 25
score on a scale | 0.86 (0.87) | 1.32 (0.54)

3. Primary Outcome: Change in Self-reported Interpretation Bias as Measured by the Children's Automatic Thoughts Scale (CATS)
Description: The Children's Automatic Thoughts Scale is a youth self-report questionnaire which assesses presence and frequency of a variety of anxious thoughts from domains of: physical threat, social threat, personal failure, and anxious hostility. Total scores range from 0 to 160, with higher scores indicating more threat interpretation bias. Higher scores indicate "worse" outcome, or that youth self-report that they have more threatening thoughts and/or threatening thoughts at higher frequency; lower scores indicate "better" outcome or that youth self-report fewer threatening thoughts and/or threatening thoughts at lower frequency.
Time Frame: 6 weeks; post-intervention time point
Population: The outcome measures data below provides the measure endorsed at the post-treatment (6 weeks) endpoint, and does not reflect the complex linear, quadratic, and piecewise models of change for analyses in Aims 1 and 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Number analyzed (Participants) | 25 | 25
score on a scale | 6.52 (10.22) | 19.00 (16.47)

4. Secondary Outcome: Number of Trainings Completed of 16 Intended Sessions
Description: This outcome is related to the "feasibility of CBM-I" aim. The number of CBM-I/ICC trainings completed of 16 intended sessions. Theoretically, completion of more training sessions is better and indicates that youth received a higher "dose" of training.
Time Frame: 6 weeks; post-intervention time point
Population: The average number of 16 possible CBM-I/ICC trainings completed per group. Note that this number averages (i.e., Mean score) across all participants in the randomized group. Two participants (siblings) dropped from CBM-I following the second training session due to an unrelated medical emergency and hospitalization, and one participant was removed from the ICC group following randomization and before completion of any trainings due to participant not being eligible for study participation.
Measure: Mean (Standard Deviation); unit: number of 16 trainings completed
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Number analyzed (Participants) | 23 | 24
number of 16 trainings completed | 16 (0) | 15.83 (0.82)

5. Secondary Outcome: Participant/Parent Acceptability Questionnaire (PAQ)
Description: The Participant Acceptability Questionnaire is a 10-item youth and parent report questionnaire, accompanied by an exit interview, that assesses burden (travel, boredom), credibility of computerized intervention techniques, and youth comprehension of the intervention. Parents and youth completed the PAQ separately.
Time Frame: 6 weeks
Population: The PAQ is scored on a scale from 0 to 50, with higher scores indicating higher acceptability. Scores of 30-39 indicate moderate acceptability and scores of 40-50 indicate high acceptability.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
Number analyzed (Participants) | 23 | 24
score on a scale
  Parent PAQ | 47.25 (5.17) | 42.91 (4.03)
  Youth PAQ | 38.61 (8.03) | 33.87 (8.41)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from study visit 2 (post-randomization and post-eligibility determination at Visit 1), and weekly through week 6 of study participation.
Description: Adverse events were queried at each study visit starting study visit 2 after participants were enrolled. The independent evaluator queried youth and caregiver separately about potential adverse events using a table provided by the NIMH CREST program. Nearly all adverse events were either COVID related (e.g., participant was exposed to or had COVID transmission from their daily life activities) or cold/flu related.
Arm/Group | Cognitive Bias Modification for Interpretations (CBM-I) | Interpretation Control Condition (ICC)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/25 | 4/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Bias Modification for Interpretations (CBM-I) (N=25) | Interpretation Control Condition (ICC) (N=25)
COVID, cold, flu, other illness (General disorders) | 5 (25) | 4 (25)

LIMITATIONS AND CAVEATS:
The trial was funded in January 2020, and recruitment scheduled to begin in April 2020. COVID shutdowns in March 2020 led to delays in initiating recruitment, continued delays in recruitment, and COVID-related illnesses that led to enrolled participants rescheduling their in-person study visits beyond the initially scheduled 6 weeks of study participation for the first 2.5 years of recruitment. Our analytic method allows for controlling for number of days in study to address this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04245501/Prot_SAP_000.pdf